CLINICAL TRIAL: NCT00003755
Title: Phase I Study of R031-7453, a Novell Cell Cycle Inhibitor, Administered as Escalating Oral Doses in Adults With Solid Tumors: 4-Day Schedule
Brief Title: Ro 31-7453 in Treating Patients With Locally Advanced or Metastatic Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 98-099; CDR0000066879 (Registry Identifier: PDQ (Physician Data Query)); ROCHE-NO15857A; NCI-G99-1499
Record Dates: First submitted 1999-11-01; First posted 2004-06-03 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Drug: MKC-1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of Ro 31-7453 in treating patients who have locally advanced or metastatic solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of Ro 31-7453 in patients with solid tumors. II. Determine the toxicity of Ro 31-7453 in this patient population. III. Evaluate the pharmacokinetics and major metabolites of Ro 31-7453 in these patients. IV. Assess any antitumor activity of Ro 31-7453 in these patients.

OUTLINE: This is a dose escalation study. Patients are treated on one of two treatment arms. In the first stage, cohorts of 1 patient each on arm I receive oral Ro 31-7453 twice daily on days 1-4, and cohorts of 1 patient each on arm II receive oral Ro 31-7453 once daily on days 1-4 at two dose levels higher than for arm I. Dose escalation ceases for each arm with the first instance of dose limiting toxicity (DLT). Two additional patients are entered at the stopping dose for each arm. If no further DLT occurs, the study proceeds to the second stage. In the second stage, dose escalation continues in increments of one dose level for each dosing schedule (arms I and II). Cohorts of 3-6 patients receive escalating doses of Ro 31-7453 in the absence of DLT. If 2 of 6 patients experience DLT at a dose level, escalation ceases and the maximum tolerated dose is defined as the previous dose level. Treatment continues every 3 weeks for 8 courses in the absence of disease progression or unacceptable toxicity. After completion of the 8 courses, patients may continue treatment until disease progression at the discretion of the investigator and the study sponsor. Patients are followed at 4 weeks.

PROJECTED ACCRUAL: A maximum of 40 patients will be accrued for this study over 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed locally advanced and/or metastatic solid tumors for which no standard therapy is available No known CNS metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: At least 12 weeks Hematopoietic: Hemoglobin at least 9 g/dL WBC at least 3,000/mm3 Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) ALT and/or AST no greater than 2.5 times ULN (no greater than 4.0 times ULN if liver or bone metastasis present) Alkaline phosphatase no greater than 2.5 times ULN (no greater than 4.0 times ULN if liver or bone metastasis present) Renal: Creatinine no greater than 1.5 times ULN OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Fertile patients must use effective contraception No history of other serious medical conditions

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks since mitomycin or nitrosoureas) Endocrine therapy: At least 4 weeks since prior hormonal therapy Concurrent antiandrogen therapy allowed Radiotherapy: At least 4 weeks since prior extended field radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1998-10; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Soignet, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States